CLINICAL TRIAL: NCT07036744
Title: When The Mirror Is Wrong: A Multi-Method Efficacy Study Of An Acceptance And Compassion-Based Group Intervention For Body Dysmorphia
Brief Title: When The Mirror Is Wrong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Maria Coimbra, Clinical Psychologist; PhD Fellow, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.12380.BD; 2022.12380.BD (Other Grant/Funding Number: FUNDAÇÃO PARA A CIÊNCIA E TECNOLOGIA)
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Body Dysmorphic Disorder
Keywords: Body Dysmorphic Disorder; Dysmorphic Concern; Acceptance and Commitment Therapy; Compassion; Psychological Flexibility; online group intervention
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Intervention Model Description: This project will follow a longitudinal design. Adults presenting with BDD symptomatology will be randomly allocated to the Control Group (no intervention; n ≥ 8) or to the Intervention Group (Mind-over-Mirror group intervention; n ≥ 8).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants who present significant Body Dysmorphia Symptomatology, as assessed during the screening stage (n ≥ 8) not subjected to any clinical psychology intervention during the period of the current trial. Participants in this group will be assessed at baseline, post-intervention [immediately after session 8], and at the 3-month follow-up. They will also be asked to monitor their weekly symptoms through a short self-report assessment.
- Intervention group (Experimental): Participants who present significant Body Dysmorphia Symptomatology, as assessed during the screening stage (n ≥ 8) subjected to an online manualized group psychological intervention - Mind-over-Mirror. This group will be assessed at baseline, post-intervention [immediately after session 8], and at the 3-month follow-up). They will also be asked to monitor their weekly symptoms through a short self-report assessment.
  Interventions: Behavioral: MIND-over-MIRROR

INTERVENTIONS:
Behavioral: MIND-over-MIRROR — An eight session (plus one follow-up booster session) on Acceptance and Commitment Therapy (ACT) with compassion developed specifically for BDD, in a group setting and applied remotely or in hybrid format.
  Arms: Intervention group

SUMMARY:
Body Dysmorphic Disorder (BDD) is a severe psychiatric condition characterized by persistent and intrusive preoccupations with perceived flaws in physical appearance, which are typically unnoticeable or appear minor to others. BDD is associated with significant psychological distress, functional impairment, and reduced quality of life. Despite its prevalence and clinical severity, BDD remains frequently underdiagnosed and misdiagnosed. While Cognitive Behavioural Therapy (CBT) and Selective Serotonin Reuptake Inhibitors (SSRIs) are currently considered standard treatments, emerging evidence suggests that third-wave psychotherapies, such as Acceptance and Commitment Therapy (ACT) and Compassion-Focused Interventions, may offer additional benefits.

This project aims to advance clinical care and scientific understanding of BDD by developing, implementing, and evaluating the preliminary efficacy of MIND-over-MIRROR-a novel group-based psychological intervention integrating ACT and compassion-based strategies for individuals exhibiting high levels of BDD symptomatology. The intervention consists of eight weekly sessions and one follow-up booster session, delivered in an online or hybrid format. A randomized feasibility study will be conducted to examine the intervention's acceptability, practicality, and preliminary clinical efficacy in adults aged 18 to 65 years. A multi-method assessment framework will be employed, with self-report measures collected at baseline, post-intervention, and 3-month follow-up. Additionally, participants from experimental and control groups will report on their weekly BDD symptomatology.

Participants in the intervention group who consent will also undergo computerized behavioural tasks and functional neuroimaging using functional near-infrared spectroscopy (fNIRS) to explore neural and cognitive correlates of treatment outcomes. Improvements are expected in core clinical outcomes, including BDD symptom severity, and it is hypothesized that changes in targeted psychological processes (e.g., self-compassion) will mediate these effects. This study will contribute novel and clinically relevant data regarding the feasibility and potential effectiveness of contextual behavioural therapies for BDD, with implications for both research and practice.

DETAILED DESCRIPTION:
Body dysmorphic disorder (BDD) is a mental disorder described by an excessive preoccupation or obsession with a perceived defect or imperfection in one's physical appearance or body functionality that is either imperceptible or barely noticeable by others, as defined in the DSM-5. While general appearance concerns are normal, in BDD these concerns are taken to the extreme and have a great impact on the individual's daily functioning and quality of life. To match diagnostic criteria, individuals must also engage in repetitive activities/compulsions (e.g., mirror checking, skin plucking, and excessive grooming). BDD is also known to be associated with poor cognitive flexibility, impulsivity, and affective processing, showing specific neural correlates. BDD is a serious mental condition that can cause a great deal of distress. However, BDD has been globally overlooked and in Portugal, before the current project, screening or assessment measures had not yet been validated, and no specialised treatment options are currently available. BDD has long been underdiagnosed, since it usually involves a lack of insight, delusional beliefs, and is highly associated with shame and severe body-image problems, leading to symptom concealment.

In the last decades, pharmacological (Serotonin reuptake inhibitors) and Cognitive Behavioural Therapy (CBT) interventions have been successfully developed for the treatment of BDD, but with some limitations, specifically regarding relapse rates. More recently, 3rd generation interventions, such as Acceptance and Compassion-based therapy, have shown promising results in BDD-related disorders (e.g., obsessive-compulsive and eating disorders) as well as with non-clinical samples (e.g., body dissatisfaction).

Despite its promising results, the application of 3rd generation interventions in BDD is still limited. So far, only pilot studies have tested such interventions in adults with BDD symptomatology. In addition, several authors have recommended integrating compassion in the treatment of BDD, working to increase and specifically target shame and self-criticism, but no studies test the efficacy of compassion skills/strategies for BDD. Our hypothesis is that by targeting specific processes involved in the development of BDD, not only will symptoms improve, but overall quality of life and relapse rates will be positively impacted. This project aims to foster the assessment and treatment of BDD while contributing to the progress of 3rd generation interventions.

Thus, we will adapt, implement, and investigate the feasibility and preliminary efficacy of the online version of the Mind-over-Mirror, an innovative programme, which combines ACT and compassion-strategies, to be delivered in group format to individuals presenting BDD symptomatology. The programme's feasibility and preliminary efficacy will be evaluated within a parallel arm study comparing against a control condition/waiting list (individuals with BDD symptomatology who will not receive any type of psychological intervention during the course of the trial). A longitudinal and multi-methods outcomes approach will be implemented (primary outcome: BDD symptomatology; secondary outcomes: general mental health [depression] and ACT, and compassion-related psychological processes [self-compassion, body-specific and general psychological flexibility, and self-criticism]; other non-mandatory and exploratory outcomes: cognitive functioning [Emotional Stroop Task and Emotion Recognition Task] and associated brain activity changes using functional Near-Infrared Spectroscopy (fNIRS). All participants will be assessed at three moments (baseline, post-intervention and 3-month follow-up), as well as report weekly BDD symptomatology.

All procedures inherent to this project were approved by the Ethics Committee of the Faculty of Psychology and Educational Sciences, University of Coimbra. Informed consent from each participant was required prior to any data collection. The voluntary, confidential and pseudo-anonymised nature of the project was clearly explained, as well as the option to decline or withdraw at any moment without any negative consequence.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years;
* Fluent Portuguese speakers;
* Over the cut-off score for the AAI (≥ 21) and the DCQ (≥ 9);

Exclusion Criteria:

* Pregnant;
* If medicated, not stabilized for at least 2 months
* Currently under other clinical psychology intervention;
* Current suicidal ideation;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Appearance Anxiety Inventory | Baseline, Weeks 1-8, 3-month follow-up
  The Appearance Anxiety Inventory (AAI) is a brief 10 item self-report scale that assesses the cognitive and behavioral aspects of BDD in particular. This scale was specifically developed by the original authors as both an outcome and process measure, since it can track changes in these processes and behaviors during treatment. Besides its global score, the AAI includes three subscales: threat monitoring, camouflaging, and avoidance. Each item is scored on a 4-point scale ranging from not at all (0) to much more than most people (3). A score equal or above 21 is considered high risk body image anxiety and/or Body Dysmorphic Disorder.
Dysmorphic Concern Questionnaire | Baseline, Week 8, 3-month follow-up
  The DCQ measures a person's degree of dysmorphic concern (i.e., the excessive preoccupation or concern with a perceived minor defect in one's physical appearance). This is a self-report measure with seven items, reporting on cognitive and behavioural aspects of dysmorphic concern. Each item is phrased with the question, "Have you ever…?" (e.g., "…been very concerned about some aspect of your physical appearance"). Each item is scored on a 4-point scale ranging from not at all (0) to much more than most people (3).

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 | Baseline, Week 8, 3-month follow-up
  : The PHQ-9 is a brief nine-item questionnaire used to screen for the severity of depression in adults. It's based on DSM-IV criteria for major depressive disorder and assesses symptoms like depressed mood, loss of interest, fatigue, and suicidal ideation. All items are rated on a four-point scale from not at all (0) to nearly every day (3).
Change in the Multidimensional Psychological Flexibility Inventory - 24 | Baseline, Week 8, 3-month follow-up
  The MPFI-24 is a 24-item self-report scale for the assessment of psychological flexibility/inflexibility, comprised by 12 subscales, representing psychological flexibility (i.e., Acceptance, Present Moment Awareness, Self as Context, Defusion, Values, Committed Action) and psychological inflexibility (i.e., Experiential Avoidance, Lack of Contact with the Present Moment, Self as Content, Fusion, Lack of Contact with Values, Inaction). Items (e.g., "I opened myself to all of my feelings, the good and the bad") are answered on a 6-point Likert scale (ranging from 1 = 'never true' to 6 = 'always true') reporting to the previous 2 weeks. The scores of the 6 flexibility and 6 inflexibility subscales can be averaged to create a composite score representing global flexibility and inflexibility, respectively. Previous psychometric information indicates good to excellent internal consistency values.
Self-compassion Scale | Baseline, Week 8, Follow-Up 3 Months
  The SCS is a 26-item self-report questionnaire that measures six components of self-compassion: self-kindness (five items); self-judgment (five items); common humanity (four items); isolation (four items); mindfulness (four items); and overidentification (four items). Mean scores on the six subscales can be averaged (after reverse-coding negative items) to create an overall self-compassion score. Items are rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always), with good psychometric properties.
Psychological Flexibility for Body Image | Baseline, Week 8, Follow-Up 3 Months
  The Psy-Flex-BI assesses body image-related psychological flexibility. Just like the Psy-Flex, a general psychological flexibility measure, it includes all six skills assumed to comprise psychological flexibility according to ACT theory. This scale is a 6-item measure (e.g., I can look at hindering thoughts regarding my physical appearance from a distance without letting them control me.), and items are rated on a scale from 5 ("very often") to 1 ("very rarely"). The scale was developed under the current project and has presented great psychometric properties.
Forms of Self-criticizing/Attacking and Self-reassuring Scale | Baseline, Week 8, Follow-Up 3 Months
  The FSCRS is a 22-item self-report questionnaire that measures how participants typically think and react in situations where things go wrong. The scale comprises three subscales that assess two forms of self-criticism (Inadequate Self and Hated Self) and the ability to self-soothe (Reassured Self). Participants are asked to respond according to a 5-point Likert scale ranging from (0) Not at all like me to (4) Extremely like me. The scale has consistently showed good psychometric properties.

OTHER OUTCOMES:
Emotion Recognition Task | Baseline and Follow-Up 3 Months
  The Emotion Recognition Task measures the ability to identify five basic emotions (happiness, sadness, anger, fear, disgust) in facial expressions along a continuum. A neutral condition was also included. For this study, brief videos (2s) depicting different facial expressions of real individuals were selected from the FACES database (Ebner et al., 2010). Each video is displayed on the screen, one at a time, and then the participant must select which emotion the face displayed from the 5 available options. The outcome measures for ERT cover percentage and number of correct or incorrect answers and overall response latencies. While completing this task, neuroimaging data will also be collected using fNIRS.
Emotional Stroop task | Baseline and Follow-Up 3 Months
  This task measures information processing for assessing emotions. The emotional Stroop task works by examining the response time of the participant to name colours of words presented to them. For this study, experimental stimuli were five 10-word lists developed in line with the following categories: (a) BDD-positive, (b) BDD-negative, (c) general positive, (d) general negative, and (e) neutral. Each word is displayed on the screen, one at a time, in a randomised colour (red, green, blue, and yellow) and the participant is asked to select the keyboard key corresponding to the word's colour, ignoring the word's meaning. The outcome measures for this task cover percentage and number of correct or incorrect answers, and overall response latencies. While completing this task, neuroimaging data will also be collected using fNIRS.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Coimbra, MSc, Principal Investigator — CINEICC, Faculty of Psychology and Educational Sciences, University of Coimbra; Cláudia Ferreira, PhD, Principal Investigator — CINEICC, Faculty of Psychology and Educational Sciences, University of Coimbra; Ana Ganho-Ávila, Ph.D., Principal Investigator — CINEICC, Faculty of Psychology and Educational Sciences, University of Coimbra
Locations (1):
- CINEICC, Faculty of Psychology and Educational Sciences of the University of Coimbra, Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared in order to protect participant confidentiality and in accordance with data protection regulations.